CLINICAL TRIAL: NCT00069498
Title: Impact of Co-Receptor and HIV Viral Burden on Gut Mucosa
Brief Title: Effect of an Anti-Inflammatory Drug on Gut Mucosa in HIV Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: K24AI001610-03 (NIH); K24AI001610-03 (NIH)
Record Dates: First submitted 2003-09-26; First posted 2003-09-30 (Estimated); Last update posted 2007-05-25 (Estimated); Status verified 2006-07

CONDITIONS: HIV Infections
Keywords: Mucosa; Inflammation; Tissue Viral Load; Anti-inflammatory; HIV-related diarrhea; Mucosal Inflammation; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Inflammation; Mucositis | interventions — Mesalamine

INTERVENTIONS:
Drug: 5-aminosalicylic acid

SUMMARY:
The lining of the gastrointestinal tract contains specialized lymphoid tissue that is part of the immune system. Like other parts of the immune system, HIV attacks this lymphoid tissue. This study will evaluate the effect of an anti-inflammatory drug on the lymphoid tissue in the gastrointestinal tracts of people with HIV.

DETAILED DESCRIPTION:
The gastrointestinal tract is the body's largest lymphoid organ. Because it contains significant numbers of activated memory T lymphocytes, it is a prime site for HIV infection and amplification. Mucosal T cells are extremely vulnerable to HIV infection due, in part, to a marked increase in CCR5 co-receptors. Understanding the impact of HIV on the gastrointestinal-associated lymphoid tissue (GALT) is essential and may provide insight into the profound drop in mucosal lymphocytes during early infection, persistence of tissue viral replication in the setting of undetectable plasma viral activity, and compartmentalization of HIV.

Pre-clinical studies have demonstrated that the mucosal compartment in HIV uninfected individuals is characterized by features which enhance vulnerability to HIV infection compared to blood. Once infected, the mucosal response to HIV is inflammation. This study will further evaluate the inflammatory response of mucosal tissue to HIV by examining the effect of the anti-inflammatory drug 5-aminosalicylic acid (5-ASA) on the gut mucosa.

Participants in this study will be randomly assigned to receive either 5-ASA or placebo. Participants will be enrolled in the study for 8 weeks; participants may then elect to continue on 5-ASA for an additional 16 weeks. Participants will have four screening visits in the month prior to beginning the study and four study visits during the 8-week study. Assessments will include medical interviews and physical exams, sigmoidoscopy with mucosal biopsy, and blood tests.

ELIGIBILITY:
Inclusion Criteria

* HIV infected
* Stable plasma viral load between 500 and 100,000 copies/ml for 3 months prior to study entry
* Stable antiretroviral therapy for at least 3 months prior to study entry
* CD4 cell count greater than or equal to 200 cells/mm3
* Mucosal viral RNA greater than or equal to 100 copies/microg total RNA within 2 weeks of study entry

Exclusion Criteria

* Allergy or intolerance to salicylates
* Gastrointestinal tract infection causing diarrhea or colonic inflammation
* Renal or hepatic disease
* Current opportunistic infection
* History of extensive small bowel resection (greater than 1/2 the length of the small intestine)
* History of intestinal mucosal disease (except HIV)
* Chronic, regular use of aspirin and/or anti-inflammatory agents within 7 weeks prior to study entry
* Oral, topical, or rectal steroids or 5-ASA within 3 months prior to study entry
* Certain laboratory abnormalities
* Significant neuropsychiatric symptoms that in the opinion of the study official could impact the conduct or outcome of the study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14
Dates: Start 1999-10

PRIMARY OUTCOMES:
Safety of 4.8 g/day 5-ASA in HIV infected patients with detectable viral load

SECONDARY OUTCOMES:
Time/trend decrease in mucosal viral RNA load and plasma viral RNA load, compared to placebo
reduction in cellular infiltration in treated patients versus those taking placebo
change in inflammation, as measured by tissue destruction
reduction in soluble inflammation (RANTES), CCR5 expression, and cellular infiltration of CD8
changes in certain activation markers in gut

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. Anton, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- David Geffen School of Medicine at UCLA, Los Angeles, California, United States